CLINICAL TRIAL: NCT01478087
Title: Pilot Study of Immunoadsorption Therapy for Patients With Chronic Non-Ischemic Dilated Cardiomyopathy
Brief Title: Immunoadsorption Therapy for Patients With Non-Ischemic Dilated Cardiomyopathy (DCM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated due to business reasons
Sponsor: Asahi Kasei Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMA-2011DCM Pilot Study
Record Dates: First submitted 2011-11-07; First posted 2011-11-23 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Cardiomyopathy, Dilated
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mysorba(single-arm) (Other)
  Interventions: Device: Mysorba

INTERVENTIONS:
Device: Mysorba — Subjects will undergo one cycle of five immunoadsorption (IA) treatment sessions over two weeks.

SUMMARY:
The purpose of this study is to evaluate the clinical safety and feasibility of Mysorba in patients with chronic non-ischemic dilated cardiomyopathy (DCM).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older.
2. Subject has provided written informed consent.
3. Subject has been classified as NYHA Class II or III.
4. Subject has been diagnosed with chronic non-ischemic dilated cardiomyopathy, defined as left ventricular ejection fraction (LVEF) < 40% and left ventricular end diastolic dimensions (LVEDd) > 55 millimeters (mm) or LVEDd/BSA > 3.0 cm/m2.
5. Subject was diagnosed with non-ischemic dilated cardiomyopathy ≥ 6 months and ≤ 5 years prior to screening visit.
6. Subject is on stable optimal medical therapy, consisting of ACE inhibitor (or ARB), β-blocker, and diuretic, for heart failure for at least 3 months
7. Subject and physician agree to switch subject from ACE inhibitors to ARB for the treatment duration.

Exclusion Criteria:

1. Subject has been classified as NYHA Class I or IV
2. Subject is currently pregnant, lactating, or of child-bearing potential and not taking adequate birth control as assessed by Investigator.
3. Subject is HBV, HCV or HIV positive.
4. Subject has anemia, defined as hemoglobin < 10.0 g/dL.
5. Subject has compromised renal function as reflected by a serum creatinine level >3.0 mg/dL or eGFR <30 mL/min or is currently on dialysis.
6. Subject has compromised hepatic function as measured by SGPT (ALT) or SGOT (AST) > three (3) times the upper limit of normal.
7. Subject had acute myocarditis ≤ 3 months prior to screening visit.
8. Subject has a history of diameter stenosis >70% of at least one major coronary artery, as determined by angiography or CTA obtained within the previous 5 years.
9. Subject is on immunosuppressive or immunomodulation therapy: intravenous (IV), intramuscular (IM), or oral.
10. Subject has a history of the following pre-existing heart disease:

    * myocardial infarction (MI), percutaneous coronary intervention (PCI), or coronary artery bypass graft (CABG)
    * valvular heart disease requiring repair, replacement, or balloon valvuloplasty
    * hypertrophic/restrictive cardiomyopathy or constrictive pericarditis
11. Subject is currently participating in, or ≤ 6 months prior to screening visit has participated in, an investigational study of a new drug, biologic, or device.
12. Subject has left ventricular noncompaction.
13. Subject has a left ventricular assist device (LVAD).
14. Subject has received a heart transplant.
15. Subject has DCM due to any of the following:

    * amyloidosis
    * sarcoidosis
    * connective tissue disease
    * peripartum cardiomyopathy
    * alcoholism
    * endocrine dysfunction as the primary cause of DCM
    * prior illicit drug use which the investigator feels as likely cause for the cardiomyopathy
    * hereditary and familial conditions (such as genetic dilated cardiomyopathy, familial storage disease, Heredofamilial neurologic and neuromuscular diseases)
16. Subject has undergone cardiac resynchronization therapy ≤ 6 months prior to screening visit.
17. Subject is unable to take ARB in place of ACE inhibitors.
18. Subject has a history of stroke ≤ 3 months prior to screening visit.
19. Subject currently has severe systemic infection requiring treatment with antibiotics.
20. Subject currently has hemodynamic instability defined as systolic blood pressure < 90 mm Hg without afterload reduction, or cardiogenic shock, or the need for inotropic support or intra-aortic balloon pump.
21. Subject has previously undergone immunosuppressive or immunomodulation therapy.
22. Subject has known hypersensitivity or contraindication to heparin including history of heparin induced thrombocytopenia (HIT).
23. Subject has history of drug or alcohol abuse or is currently abusing alcohol or drugs.
24. Subject has active malignancy or tumor, or other non-cardiac medical condition, which causes life expectancy to be less than one year.
25. History of neutropenia (WBC < 3,000/mm3), coagulopathy, or thrombocytopenia (platelet count < 100,000/μL) that has not resolved or has required treatment in the past 6 months.
26. Subject weighs less than 40 kg (88 lbs).
27. Subject requires major elective procedures (AHA-defined intermediate to high risk surgery) within 6 months post-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Winters, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First site open to enrollment : November 3, 2011 Study terminated: March 22, 2012
Pre-assignment Details: Three (3) subjects enrolled, 2 completed treatment through six-month follow up. One (1) subject terminated participation prior to treatment due to sponsor stopping the study.
Groups:
- IA Treatment: The Mysorba device is an immunoadsorbent column. : Subjects will undergo one cycle of five immunoadsorption (IA) treatment sessions over two weeks.
Period: Overall Study
Arm/Group | IA Treatment
Started | 3
Completed | 2
Not Completed | 1
Not completed — due to sponsor closing study | 1

BASELINE CHARACTERISTICS:
Arm/Group | IA Treatment
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54.0 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Procedure Related Serious Adverse Events (SAE) at 30 Days Post-treatment.
Time Frame: 30 Days Post Treatment
Measure: Number; unit: percentage of procedure related SAE
Arm/Group | IA Treatment
Number analyzed (Participants) | 2
percentage of procedure related SAE | 0

2. Primary Outcome: Rate of Device Related Serious Adverse Events (SAE) at 30 Days Post-treatment.
Time Frame: 30 days post-treatment
Measure: Number; unit: percentage of device related SAE
Arm/Group | IA Treatment
Number analyzed (Participants) | 2
percentage of device related SAE | 0

ADVERSE EVENTS:
Arm/Group | IA Treatment
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IA Treatment (N=3)
pulse drop (Investigations) | 1 (2)
PVC'S (Cardiac disorders) | 1 (1)
flushing (Vascular disorders) | 1 (2)
hematoma (Vascular disorders) | 1 (1)
dizzy (Nervous system disorders) | 1 (4)
loss of vascular access (Injury, poisoning and procedural complications) | 1 (1)
elevated INR (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall provide the sponsor with a copy of any proposed publication for review at least 60 days prior to submission to a publisher. The sponsor may request that any confidential information or intellectual property contained be removed, redacted, or modified. If the PI do not agree to such deletion or modification, they shall notify the sponsor and agree to postpone such submission for an additional 60 days to allow sponsor to file the appropriate applications or seek protective remedies.